CLINICAL TRIAL: NCT02148692
Title: Protective Ventilation With Higher Versus Lower PEEP During General Anesthesia for Surgery in Obese Patients
Acronym: PROBESE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ANE-PROBESE
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Morbid Obesity; Surgery; General Anesthesia
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Higher PEEP (Experimental): PEEP of 12 cmH2O or higher and lung recruitment maneuvers
  Interventions: Procedure: Higher PEEP
- Lower PEEP (Active Comparator): PEEP of 4 cmH2O without lung recruitment maneuvers
  Interventions: Procedure: Lower PEEP

INTERVENTIONS:
Procedure: Higher PEEP
  Arms: Higher PEEP
Procedure: Lower PEEP
  Arms: Lower PEEP

SUMMARY:
Postoperative respiratory failure, particularly after surgery under general anesthesia, adds to the morbidity and mortality of surgical patients. Anesthesiologists inconsistently use positive end-expiratory pressure (PEEP) and recruitment maneuvers in the hope that this may improve oxygenation and protect against postoperative pulmonary complications (PPCs), especially in obese patients. While anesthesiologists tend to use PEEP higher than in non-obese patients. While it is uncertain whether a strategy that uses higher levels of PEEP with recruitment maneuvers truly prevents PPCs in these patients, use of higher levels of PEEP with recruitment maneuvers could compromise intra-operative hemodynamics.

The investigators aim to compare a ventilation strategy using higher levels of PEEP with recruitment maneuvers with one using lower levels of PEEP without recruitment maneuvers in obese patients at an intermediate-to-high risk for PPCs.

We hypothesize that an intra-operative ventilation strategy using higher levels of PEEP and recruitment maneuvers, as compared to ventilation with lower levels of PEEP without recruitment maneuvers, prevents PPCs in obese patients at an intermediate-to-high risk for PPC.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for open or laparoscopic surgery under general anesthesia
* Intermediate-to-high risk for PPCs following surgery, according to the ARISCAT risk score (≥ 26)
* BMI ≥ 35 kg/m2
* Expected duration of surgery ≥ 2 h

Exclusion Criteria:

* Age < 18 years
* Previous lung surgery (any)
* Persistent hemodynamic instability, intractable shock (considered hemodynamically unsuitable for the study by the patient's managing physician)
* History of previous severe chronic obstructive pulmonary disease (COPD) (non-invasive ventilation and/or oxygen therapy at home, repeated systemic corticosteroid therapy for acute exacerbations of COPD)
* Recent immunosuppressive medication (patients receiving chemotherapy or radiation therapy up to two months prior to surgery)
* Severe cardiac disease (New York Heart Association class III or IV, acute coronary syndrome or persistent ventricular tachyarrhythmias)
* Invasive mechanical ventilation longer than 30 minutes (e.g., general anesthesia for surgery) within last 30 days
* Pregnancy (excluded by anamneses and/or laboratory analysis)
* Prevalent acute respiratory distress syndrome expected to require prolonged postoperative mechanical ventilation
* Severe pulmonary arterial hypertension, defined as systolic pulmonary artery pressure > 40 mmHg
* Intracranial injury or tumor
* Neuromuscular disease (any)
* Need for intraoperative prone or lateral decubitus position
* Need for one-lung ventilation
* Cardiac surgery
* Neurosurgery
* Planned reintubation following surgery
* Enrolled in other interventional study or refusal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2013 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | Five postoperative days
Hospital-free days at day 90 | 90 postoperative days
Mortality at day 90 | 90 postoperative days
Postoperative extra-pulmonary complications | Five postoperative days
Postoperative wound healing | Five postoperative days

SECONDARY OUTCOMES:
Intra-operative complications | Surgery period
  complications related to the ventilation strategy (for example: de-saturation, defined as SpO2 ≤ 92%, for > 1 min; hypotension during recruitment maneuvers, as defined by systolic arterial pressure < 90 mmHg for > 2 min)
Need for postoperative ventilatory support | Five postoperative days
  invasive or non-invasive ventilation
Unexpected need for ICU admission or ICU readmission within 30 days | Five postoperative days
Need for hospital readmission within 30 days | 30 postoperative days

CONTACTS AND LOCATIONS:
Locations (24):
- United States (2):
  - Massachusetts General Hospital, Harvard University, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
- Medical University, Vienna, Austria
- Belgium (2):
  - AZ Sint Jan Brugge-Oostende AV, Bruges
  - Ghent University Hospital, Ghent
- ABC Medical School, São Paulo, Brazil
- Saint Michael's Hospital, University of Toronto, Toronto, Canada
- Saint Eloi University Hospital, Montpellier, France
- Germany (4):
  - Department of Anesthesiology and Intensive Care, University Hospital Carl Gustav Carus, Dresden, Saxony
  - University of Aachen, Aachen
  - University of Bonn, Bonn
  - University of Leipzig, Leipzig
- Semmelweis Egyetem, Budapest, Hungary
- Tel Aviv Medical Center, Tel Aviv, Israel
- Italy (4):
  - University of Foggia, Foggia
  - University of Genoa, Genoa
  - Città della Salute e della Scienza, Turin
  - University of Insubria, Varese
- Academic Medical Center, University of Amsterdam, Amsterdam, Netherlands
- Hospital Universitari Germans Trias I Pujol, Barcelona, Spain
- University Hospital Uppsala, Uppsala, Sweden
- Hôpitaux Universitaires de Genève, Geneva, Switzerland
- University of Istanbul, Istanbul, Turkey (Türkiye)
- Sheffield Teaching Hospitals, Sheffield, United Kingdom

REFERENCES:
- [Derived] Bluth T, Rivas E, Lopez-Baamonde M, Sanahuja JM, Lopez-Hernandez A, Balust J, Weingarten TN, Girrbach F, Simon P, Wrigge H, Wittenstein J, Birr K, Teichmann R, Huhle R, Melchior N, Vivona L, Koch T, Ramakrishna H, Brull S, Serpa Neto A, Schultz MJ, Sprung J, Scharffenberg M, Gama de Abreu M; PROBESE-investigators; Protective Ventilation Network, and the Clinical Trials Network of the European Society of Anaesthesiology and Intensive Care. Association of plasma biomarkers of lung injury with positive end expiratory pressure and postoperative pulmonary complications in obese surgical patients: A substudy of the PROBESE randomised controlled trial. Eur J Anaesthesiol. 2025 Sep 1;42(9):840-850. doi: 10.1097/EJA.0000000000002221. Epub 2025 Jun 20. PMID 40548583
- [Derived] Scharffenberg M, Mandelli M, Bluth T, Simonassi F, Wittenstein J, Teichmann R, Birr K, Kiss T, Ball L, Pelosi P, Schultz MJ, Gama de Abreu M, Huhle R; PROBESE-investigators; Protective Ventilation Network; Clinical Trials Network of the European Society of Anaesthesiology and Intensive Care. Respiratory mechanics and mechanical power during low vs. high positive end-expiratory pressure in obese surgical patients - A sub-study of the PROBESE randomized controlled trial. J Clin Anesth. 2024 Feb;92:111242. doi: 10.1016/j.jclinane.2023.111242. Epub 2023 Oct 12. PMID 37833194
- [Derived] Ellenberger C, Pelosi P, de Abreu MG, Wrigge H, Diaper J, Hagerman A, Adam Y, Schultz MJ, Licker M; PROBESE investigators, of the PROtective VEntilation Network (PROVEnet); Clinical Trial Network of the European Society of Anaesthesiology and Intensive Care (ESAIC). Distribution of ventilation and oxygenation in surgical obese patients ventilated with high versus low positive end-expiratory pressure: A substudy of a randomised controlled trial. Eur J Anaesthesiol. 2022 Nov 1;39(11):875-884. doi: 10.1097/EJA.0000000000001741. Epub 2022 Sep 12. PMID 36093886
- [Derived] Writing Committee for the PROBESE Collaborative Group of the PROtective VEntilation Network (PROVEnet) for the Clinical Trial Network of the European Society of Anaesthesiology; Bluth T, Serpa Neto A, Schultz MJ, Pelosi P, Gama de Abreu M; PROBESE Collaborative Group; Bluth T, Bobek I, Canet JC, Cinnella G, de Baerdemaeker L, Gama de Abreu M, Gregoretti C, Hedenstierna G, Hemmes SNT, Hiesmayr M, Hollmann MW, Jaber S, Laffey J, Licker MJ, Markstaller K, Matot I, Mills GH, Mulier JP, Pelosi P, Putensen C, Rossaint R, Schmitt J, Schultz MJ, Senturk M, Serpa Neto A, Severgnini P, Sprung J, Vidal Melo MF, Wrigge H. Effect of Intraoperative High Positive End-Expiratory Pressure (PEEP) With Recruitment Maneuvers vs Low PEEP on Postoperative Pulmonary Complications in Obese Patients: A Randomized Clinical Trial. JAMA. 2019 Jun 18;321(23):2292-2305. doi: 10.1001/jama.2019.7505. PMID 31157366
- [Derived] Bluth T, Teichmann R, Kiss T, Bobek I, Canet J, Cinnella G, De Baerdemaeker L, Gregoretti C, Hedenstierna G, Hemmes SN, Hiesmayr M, Hollmann MW, Jaber S, Laffey JG, Licker MJ, Markstaller K, Matot I, Muller G, Mills GH, Mulier JP, Putensen C, Rossaint R, Schmitt J, Senturk M, Serpa Neto A, Severgnini P, Sprung J, Vidal Melo MF, Wrigge H, Schultz MJ, Pelosi P, Gama de Abreu M; PROBESE investigators; PROtective VEntilation Network (PROVEnet); Clinical Trial Network of the European Society of Anaesthesiology (ESA). Protective intraoperative ventilation with higher versus lower levels of positive end-expiratory pressure in obese patients (PROBESE): study protocol for a randomized controlled trial. Trials. 2017 Apr 28;18(1):202. doi: 10.1186/s13063-017-1929-0. PMID 28454590